CLINICAL TRIAL: NCT00174499
Title: An Open-label Study on Nicorette Freshmint Gum, 2 MG AND 4 MG in Smokers With Visible Teeth Staining Motivated to Quit
Brief Title: A Pilot Drug Trial That Evaluates the Whitening Potential of Nicotine Gum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A6431088
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Dental Pellicle
Keywords: Tooth stain
MeSH Terms: conditions — Tooth Discoloration | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2 mg nicotine gum
  Interventions: Drug: 2 mg nicotine gum
- 2 (Experimental): 4 mg nicotine gum
  Interventions: Drug: 4 mg nicotine gum

INTERVENTIONS:
Drug: 2 mg nicotine gum — 2 mg nicotine gum
  Other Names: Nicorette Fresh Mint
  Arms: 1
Drug: 4 mg nicotine gum — 4 mg nicotine gum
  Other Names: Nicorette Fresh Mint
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate the effects on existing tooth stain of nicotine gum. The study will enroll adults who have visible tooth staining.

DETAILED DESCRIPTION:
This was a 6-week, open-label, single-center study conducted in 78 subjects who were smokers with visible staining of teeth and who were motivated to quit smoking through use of Nicorette Freshmint gum.

The subjects were assigned, per label instructions, to either Nicorette Freshmint gum 2 mg or 4 mg based on the number of cigarettes smoked per day. Subjects who smoked at least 25 or more cigarettes per day were assigned to the 4 mg gum group; those who smoked less than 25 cigarettes per day were assigned to the 2 mg gum group.

A total of 3 study visits were planned: Screening/Baseline, Week 2 and Week 6. A telephone screening prior to Baseline and the Screening/Baseline visit was performed to confirm subject eligibility. At each visit an oral examination, including a stain index measurement used to rate tooth-staining (MacPherson Modification of the Lobene Stain Index), was conducted; and smoking status and motivation to quit smoking were assessed. The safety evaluation at each visit included an oral tissue assessment in addition to assessment for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* daily smokers for at least one year
* motivated to quit smoking
* normal chewing ability
* willing to refrain from a dental prophylaxis for the duration of the study
* total extrinsic facial tooth stain score > or = to 28, according to the MacPherson Modification of the Lobene Stain Index

Exclusion Criteria:

* < 20 natural teeth
* inadequate oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to assess, by using the MacPherson modification of the Lobene Stain Index, the amount of extrinsic tooth-stain reduction from Baseline while quitting smoking using Nicorette Freshmint gum | 6 Weeks

SECONDARY OUTCOMES:
To assess reduction in tooth-staining in relation to usage of gums | 6 Weeks
To assess smoking status | 6 Weeks
To assess safety | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth A Kruse, PhD, Study Director — JJCPPW